CLINICAL TRIAL: NCT05592093
Title: An RCT Study to Investigate the Effect of Korean Red Ginseng for Middle-aged and Elderly Sub-health Population on Anti-oxidation
Brief Title: Effect of Korean Red Ginseng on Oxidation in Middle-aged and Elderly Sub-health Population
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: RenJi Hospital (Other); Beijing Obstetrics and Gynecology Hospital (Other); Foshan Fuxing Changcheng Hospital (Unknown); Nanchang Hongdu Hospital of TCM (Unknown)
Responsible Party: Principal Investigator, Hongsheng Tan, professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KRGO-2022
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy Ageing; Antioxidative Stress
Keywords: Korean Red ginseng; Healthy Ageing; Antioxidant Effect
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Intervention Model Description: A Phase 2/3 Randomized, Double-blind, Placebo-controlled, Multicenter Study of Korean red ginseng capsule Administered by taking orally in Middle-aged and Elderly Sub-health population.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KRGO group (Experimental): Korean red ginseng capsule (KRGO)marketed product in Korea donated by The Korean Society of Ginseng.
  Interventions: Drug: Korean red ginseng capsule (marketed product in Korea)
- placebo group (Placebo Comparator): Same smell, color and shape as Korean red ginseng capsule (KRGO)without herbs in capsules.
  Interventions: Drug: Korean red ginseng capsule(placebo)

INTERVENTIONS:
Drug: Korean red ginseng capsule (marketed product in Korea) — Korean red ginseng capsule (marketed product in Korea) KRGO group and placebo group were used for treatment. The random number is generated by the central randomization system. All the recruiters were divided into placebo group and KRGO group. The numbers will be assigned according to random numbers. In this study, qualified subjects were randomly assigned to the KRGO group and placebo group at a ratio of 1:1. The drug was administered for 12 weeks, 2 times a day, 3 capsules each time.
  Other Names: red ginseng
  Arms: KRGO group
Drug: Korean red ginseng capsule(placebo) — KRGO group and placebo group were used for treatment. The random number is generated by the central randomization system. All the recruiters were divided into placebo group and KRGO group.
  The numbers will be assigned according to random numbers. In this study, qualified subjects were randomly assigned to the KRGO group and placebo group at a ratio of 1:1. The drug was administered for 12 weeks, 2 times a day, 3 capsules each time.
  Other Names: placebo group
  Arms: placebo group

SUMMARY:
The objective of this study is to examine the effects and safety of Korean red ginseng capsule and placebo with middle-aged and elderly sub-health population.

DETAILED DESCRIPTION:
Processed red ginseng are non-toxic and healthy "tonics". It was recorded in medical books and Materia Medica that taking it for a long time can prolong life. The main purpose of this study is to evaluate the effect of ginseng on antioxidation and healthy aging indicators of sub-health subjects in Han Chinese population. Subjects will undergo a safety follow-up after the treatment period. Safety and efficacy will be determined by looking at a number of assessments [physical examinations, blood sampling, sub-health status evaluation questionnaire (shsq-25), etc.]. It is expected that around 900 people (at least 450 in each arm) with sub-healthy state may take part in the study. The study participants will be recruited at around 3 sites from Northern(Beijing),Central(Shanghai), Southern(Foshan and Nanchang) in China.

ELIGIBILITY:
Inclusion Criteria:

1. 40-75 years old, male or female, Han nationality;
2. There was no history of major chronic disease or clinically active disease within 3 months before the study, including any cardiovascular, cerebrovascular, lung, kidney, liver, endocrine, digestive tract, nervous system or metabolic disease; Inflammation, psychosis, AIDS, tumor or traumatic injury, etc., and the disease history that the researcher judges to have an impact on the study;
3. According to the sub-health status evaluation questionnaire (shsq-25), ≥ 35 points can be judged as sub-health;
4. Agree to have no family planning or sperm donation plan during the trial and within 6 months after the end of the trial and voluntarily take effective contraceptive measures (avoid using contraceptives);
5. Cohabitants included only one subject; Those who sign the informed consent shall fully understand the test content, process and possible adverse reactions, and be able to communicate well with the investigator.

Exclusion Criteria:

1. Those who need to take medicine (traditional Han Chinese medicine, western medicine, biological medicine) due to any major chronic disease or clinically active disease within 3 months before the study;
2. Obesity population (BMI index) (kg / m2) BMI ≥ 28KG / m2; Low body weight population (BMI index) (kg / m2) BMI < 18.5kg/m2;
3. Vegetarians within 3 months before the study;
4. Those who took other antioxidant health products within 3 months before the study (vitamin health products or supplements; zinc and selenium health products or supplements; superoxide dismutase (SOD) health products; health products containing grape seeds, lycopene, flavonoids, astaxanthin, propolis, squalene, nicotinamide nucleoside, omega-3 or omega-6, etc.);
5. Those who took (or used) microecological regulators within 3 months before the study;
6. Those who drank more than 200ml of coffee per day (converted as pure coffee) within 3 months before the study;
7. Those who are known to be allergic to red ginseng ingredients, or who have a specific history of allergy (asthma, measles, eczema, etc.), or allergic constitution (such as those who are allergic to two or more drugs, food such as milk and pollen), or who have a history of food, drug hypersensitivity or allergic reaction judged by other researchers to have clinical significance;
8. Alcoholics (drinking more than 14 standard units per week. 1 standard unit contains 14g alcohol, such as 360ml beer or 45ml spirit with 40% alcohol or 150ml wine), or those with positive breath test within 3 months before the study；
9. Those who smoked more than 10 cigarettes per day in the 3 months before the study;
10. Those who have participated in or are participating in other clinical trials within 3 months before the study;
11. The investigator considered that there were other patients who were not suitable to participate in this study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Change in malondialdehyde (MDA) after 12 weeks of treatment | 12 weeks
  To compare the change in serum MDA from baseline (week 1 to week 12) between KRGO and placebo.

SECONDARY OUTCOMES:
Change in serum lipofuscin after 12 weeks of treatment | 12 weeks
  To compare the changes in serum lipofuscin from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum protein carbonyl after 12 weeks of treatment | 12 weeks
  To compare the changes in serum protein carbonyl from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum 8-hydroxy-2'-deoxyguanosine(8-OHdG) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum 8-OHdG from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum superoxide dismutase (SOD) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum SOD from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum glutathione(GSH) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum GSH from baseline (week 1 to week 12) between KRGO and placebo.
Changes in the sub-health status evaluation questionnaire (shsq-25) after 12 weeks and 16 weeks treatment | 12 weeks # 16 weeks
  To compare the change in the sub-health status evaluation questionnaire (shsq-25) using face to face Interview for the scores from baseline (week 1 to week 12, week 12 to week 16) between KRGO and placebo (range, 0 [best] to 100 [worst]).

OTHER OUTCOMES:
Change in serum total cholesterol(TC) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum TC from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum triglyceride(TG) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum TG from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum low density lipoprotein (LDLC) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum LDLC from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum high density lipoprotein (HDLC) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum HDLC from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum apolipoproteins after 12 weeks of treatment | 12 weeks
  To compare the changes in serum apolipoprotein from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum lipoproteins after 12 weeks of treatment | 12 weeks
  To compare the changes in serum lipoprotein from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum Fasting Blood Glucose after 12 weeks of treatment | 12 weeks
  To compare the changes in Fasting Blood Glucose (FBG) from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum glycated hemoglobin ( HbA1c) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum glycated hemoglobin ( HbA1c) from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum C-reactive protein (CRP) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum CRP from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum cytokines after 12 weeks of treatment | 12 weeks
  To compare the changes in serum cytokines from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in serum immunoglobulin G (IgG) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum IgG from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in serum immunoglobulin A (IgA) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum IgA from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in serum immunoglobulin M (IgM) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum IgM from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in Peripheral Blood Mononuclear Cells after 12 weeks of treatment | 12 weeks
  To compare the changes in Peripheral Blood Mononuclear Cells from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in serum estradiol (E2) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum E2 from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum follicle stimulating hormone (FSH) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum FSH from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum luteinizing hormone (LH) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum LH from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum testosterone after 12 weeks of treatment | 12 weeks
  To compare the changes in serum testosterone from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum prolactin (PRL) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum PRL from baseline (week 1 to week 12) between KRGO and placebo.
Change in serum progesterone (P) after 12 weeks of treatment | 12 weeks
  To compare the changes in serum P from baseline (week 1 to week 12) between KRGO and placebo.
Mean change from baseline to Week 12 in Composite Clinical Indicator Score | 12 weeks
  Composite Clinical Indicator Score is a prespecified unitless composite index summarizing [cardiometabolic / vascular aging / biological aging] status. It is constructed following the principles in the OECD/JRC Handbook on Constructing Composite Indicators (theoretical framework, indicator selection, missing data handling, normalization, weighting and aggregation).
  Component indicators are prespecified and grouped into domains:
  1. Lipid/atherogenicity domain: [TG, HDL-C, LDL-C, …]
  2. Glycemic/metabolic domain: [fasting glucose, HbA1c, …]
  3. Blood pressure/vascular domain: [SBP, DBP, …]
  4. Inflammation domain: [hsCRP, …] Each component is standardized to z-scores using baseline distribution, then aggregated using [equal weights / prespecified weights / PCA-derived weights] with linear aggregation to yield a unitless Composite Clinical Indicator Score.
Change in perpheral metabolomics after 12 weeks of treatment | 12 weeks
  Peripheral venous blood will be collected at baseline (Week 1) and Week 12. Serum metabolomics will be quantified using LC-MS/MS. Metabolomics levels will be reported as normalized relative abundance. The outcome is the change from baseline to Week 12 in normalized metabolomics levels.
Change in perpheral Protein Levels after 12 weeks of treatment | 12 weeks
  Peripheral venous blood will be collected at baseline (Week 1) and Week 12. Plasma/serum proteins will be quantified using [Olink / SOMAscan / LC-MS/MS]. Protein levels will be reported as normalized relative abundance. The outcome is the change from baseline to Week 12 in normalized protein levels.
Change in perpheral Gene Expression Profile after 12 weeks of treatment | 12 weeks
  Whole blood will be collected at baseline (Week 1) and Week 12. RNA will be extracted and next-generation RNA sequencing (RNA-seq)/DNA methylation/epigenomics be performed. Gene expression will be quantified as normalized expression values and the outcome is the change from baseline to Week 12 in gene expression.
Change in Gut Microbiota 16S rRNA/shotgun metagenomic after 12 weeks of treatment | 12 weeks
  Stool samples will be collected at baseline (Week 1) and Week 12. Gut microbiota will be assessed by 16S rRNA amplicon sequencing and sequence variants (ASVs) will be derived using a standard denoising pipeline. Alpha-diversity will be summarized as the number of observed ASVs. The outcome is the change from baseline to Week 12 in observed ASVs.
Change in The Short-Form 36 physical component summary (SF-36 PCS) after 12 weeks and 16 weeks of treatment | 12 weeks # 16 weeks
  To compare the change in SF-36 PCS using Face to face Interview for the scores from baseline (week 1 to week 12， week 12 to week 16) between KRGO and placebo. (range, 0 [best] to 100 [worst])
Change in the TCM Physique Questionnaire score after 12 weeks and 16 weeks of treatment | 12 weeks # 16 weeks
  To compare the change in the TCM Physique Questionnaire using Face to face Interview for the scores from baseline (week 1 to week 12, week 12 to week 16) between KRGO and placebo (range, 0 [best] to 100 [worst]).
Change in muscle strength with hydraulic type handgrip dynamometer or spring type handgrip dynamometer after 12 weeks of treatment | 12 weeks
  To compare the change in muscle strength with hydraulic type handgrip dynamometer or spring type handgrip dynamometer from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in skeletal muscle mass index (SMI) after 12 weeks of treatment | 12 weeks
  To compare the change in SMI with spring grip from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in appendicular skeletal muscle mass (ASM) after 12 weeks of treatment | 12 weeks
  To compare the change in ASM from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in percentage body fat (PBF) after 12 weeks of treatment | 12 weeks
  To compare the change in PBF from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in body fat mass (BFM) after 12 weeks of treatment | 12 weeks
  To compare the change in BFM from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in visceral fat area (VFA) after 12 weeks of treatment | 12 weeks
  To compare the change in VFA from baseline (week 1 to week 12) between KRGO and placebo. Patients from lead trial center were selected for this study.
Change in Complete Blood Count after 12 weeks of treatment | 12 weeks
  To compare the change in Complete Blood Count from baseline (week 1 to week 12) between KRGO and placebo.
Change in Urinalysis Parameters (Urine Dipstick and Microscopy) after 12 weeks of treatment | 12 weeks
  A midstream clean-catch urine sample will be collected at Baseline (Week 1) and Week 12. Urinalysis will be performed using an automated urine dipstick analyzer and microscopic examination of urine sediment per standard clinical laboratory procedures. Parameters assessed include dipstick chemistry and microscopic sedimen. The outcome is the change from baseline to Week 12 in urinalysis results (reported in conventional laboratory units/grades as applicable by the testing laboratory).
Change in Liver Function Tests after 12 weeks of treatment | 12 weeks
  Venous blood will be collected at Baseline (Week 1) and Week 12. Liver function tests will be measured by a certified clinical laboratory using standard automated clinical chemistry analyzers (enzymatic/photometric methods as applicable). Analytes include alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma-glutamyltransferase (GGT), total bilirubin, and albumin. e.g. Results will be reported in standard units (e.g., U/L for enzymes; mg/dL or µmol/L for bilirubin; g/dL for albumin). The outcome is the change from baseline to Week 12 for each analyte.
Change in Renal Function Tests after 12 weeks of treatment | 12 weeks
  The change in renal function from Baseline (Week 1) to Week 12 will be monitored through a standard clinical laboratory profile. Venous blood will be processed by a certified facility to measure a composite of renal health indicators, including serum creatinine, BUN, and eGFR (calculated via CKD-EPI). etc. These metrics serve as a combined dataset to evaluate the subject's overall renal physiological status and filtration capacity throughout the study duration.
Change in Chinese Medicine Fire Heat Syndrome Scale after 12 weeks and 16 weeks of treatment | 12 weeks # 16 weeks
  To compare the change in Chinese Medicine Fire Heat Syndrome Scale using Face to face Interview for the scores from baseline (week 1 to week 12, week 12 to week 16) between KRGO and placebo. (range, 0 [best] to 100 [worst])
Change in participants from Baseline (Week 1) to Week 12 in physiological parameters by Huawei sports bracelet daily | Baseline (Week 1) and Week 12 (end of continuous 12-week monitoring period).
  From the basline，participants will wear a Huawei wrist-worn wearable device continuously from Baseline (Week 1) through Week 12. Physiologic signals are collected by the device sensors (e.g., PPG for heart rate/SpO2; accelerometer + PPG for sleep) and summarized by the device/app's prespecified algorithms.
  Data will be synchronized via the Huawei Innovation Platform and exported for analysis.
Change in Food Frequency Questionnaire every week of treatment | Every week during 12 weeks
  From the basline，participants will record their food frequency questionnaire (FFQ) every week by Questionnaire Star/ WJX.cn. To compore the change in FFQ of participants between KRGO and placebo every week.
Change in International Physical Activity Questionnaire every week of treatment | Every week during 12 weeks
  From the basline，participants will record their International Physical Activity Questionnaire (IPAQ) every week by Questionnaire Star/WJX.cn. To compore the change in IPAQ of participants between KRGO and placebo every week. (range, 0 [best] to 100 [worst])
Change in number of participant with abnormal ECG after 12 weeks of treatment | 12 weeks
  To compare the number of participant with abnormal ECG from baseline (week 1 to week 12) between KRGO and placebo.
Adverse Events | 12 weeks
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yaomin Hu, Professor, Study Director — RenJi Hospital; Chenghong Yin, Professor, Study Director — Beijing Obstetrics and Gynecology Hospital; Suzhen Wu, Professor, Study Director — Foshan Fuxing Changcheng Hospital
Locations (4):
- China (4):
  - Beijing Obstetrics and Gynecology Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Foshan Fuxing Changcheng Hospital, Foshan, Guangdong
  - Nanchang Hongdu Hospital of TCM, Nanchang, Jiangxi
  - Renji Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HG, Yoo SR, Park HJ, Lee NH, Shin JW, Sathyanath R, Cho JH, Son CG. Antioxidant effects of Panax ginseng C.A. Meyer in healthy subjects: a randomized, placebo-controlled clinical trial. Food Chem Toxicol. 2011 Sep;49(9):2229-35. doi: 10.1016/j.fct.2011.06.020. Epub 2011 Jun 15. PMID 21699953
- [Background] Hou W. iTRAQ-based Proteomic Analysis Reveals Anti-Aging Effects of Red Ginseng Powder on Drosophila Melanogaster and its Mechanism Studies. Jilin University, 2021. DOI:10.27162/d.cnki.gjlin.2021.000482.
- [Background] Park SK, Hyun SH, In G, Park CK, Kwak YS, Jang YJ, Kim B, Kim JH, Han CK. The antioxidant activities of Korean Red Ginseng (Panax ginseng) and ginsenosides: A systemic review through in vivo and clinical trials. J Ginseng Res. 2021 Jan;45(1):41-47. doi: 10.1016/j.jgr.2020.09.006. Epub 2020 Oct 10. PMID 33437155
- [Background] Chung TH, Kim JH, Seol SY, Kim YJ, Lee YJ. The Effects of Korean Red Ginseng on Biological Aging and Antioxidant Capacity in Postmenopausal Women: A Double-Blind Randomized Controlled Study. Nutrients. 2021 Sep 2;13(9):3090. doi: 10.3390/nu13093090. PMID 34578969
- [Background] Kim JY, Park JY, Kang HJ, Kim OY, Lee JH. Beneficial effects of Korean red ginseng on lymphocyte DNA damage, antioxidant enzyme activity, and LDL oxidation in healthy participants: a randomized, double-blind, placebo-controlled trial. Nutr J. 2012 Jul 17;11:47. doi: 10.1186/1475-2891-11-47. PMID 22805313